CLINICAL TRIAL: NCT03668509
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR1459, in Healthy Volunteers
Brief Title: Safety, Tolerability and PK/PD of SHR1459 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SHR1459-101
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers
Keywords: SHR1459; Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): oral adminstration of SHR1459, dose 1
  Interventions: Drug: SHR1459
- Cohort 2 (Experimental): oral adminstration of SHR1459, dose 2
  Interventions: Drug: SHR1459
- Cohort 3 (Experimental): oral adminstration of SHR1459, dose 3
  Interventions: Drug: SHR1459

INTERVENTIONS:
Drug: SHR1459 — oral adminstration, single dose
  Other Names: Placebo

SUMMARY:
This was a phase I, single-center, double-blind, randomized, placebo-controlled study to assess the safety, tolerability and pharmacokinetics/pharmacodynamics of the investigational medicinal product in healthy volunteers.

DETAILED DESCRIPTION:
The study originally planned to enroll 3 cohorts of 10 subjects each (N=30).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnic origin, age ≥18 and ≤45 years of age;
* BMI ≥19 and ≤26 kg/m2; Men's weight≥ 50kg, Women's weight ≥ 45kg;
* Medical history without major pathology and determined to be in good health with no clinically significant findings as assessed by the Investigator; all clinical tests of blood, urine, ECG and X-ray are within the normal range or show no clinically relevant deviations as judged by the Investigator;
* There is no birth plan during the trial and within 1 month after the completion of the trial, and the subject must agree to use one of the effective contraceptive methods;
* Able to comprehend and abide by the study restrictions, and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

* Has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
* Has a history of malignant or lymphoproliferative disorders;
* Has a history of bleeding tendency or coagulopathy (eg, uncontrolled autoimmune hemolysis and thrombocytopenic purpura, severe hematopoietic defects, gastrointestinal bleeding), or recent bleeding events;
* Has a history of stroke or intracranial hemorrhage within 6 months prior to screening;
* Has any surgery performed within 3 months prior to screening, or during the study period and within 1 month after the end of the study;
* Has a significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, immune suppressive/defective, or psychiatric disorder as determined by the Investigator;
* Has diseases affecting drug absorption, distribution, metabolism, and excretion (eg, gastrointestinal dysfunction, peptic ulcer, gastrointestinal surgery, etc);
* Has active tuberculosis by clinical symptoms, signs, laboratory tests, or X-ray examinations;
* Has infections including acute and chronic infections, local infections such as sepsis, abscesses, and opportunistic infections that were clinically significant by the investigator in the 3 months prior to screening;
* Has blood donation and donated ≥400 mL within 3 months before screening ; or received any blood product infusion; or received plasma exchange or blood cell clearance treatment;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single oral doses of SHR1459 determined by adverse events | within 4 days after single dose
  Frequency and severity of AEs and serious AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Xu qian, M.D. Ph.D, Shanghai, China